CLINICAL TRIAL: NCT07305597
Title: Effects of Virtual Reality-Assisted Pain Neuroscience Education on Chronic Nonspecific Low Back Pain: A Randomized Controlled Trial
Brief Title: Effects of Virtual Reality-Assisted Pain Neuroscience Education on Chronic Nonspecific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, İrem CANLI, Research Assistant, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23591230588=
Record Dates: First submitted 2025-12-13; First posted 2025-12-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Chronic Non-Specific Low Back Pain
Keywords: chronic non-spesific low back pain; virtual reality; pain neuroscience education

STUDY DESIGN:
Intervention Model Description: Randomized dontrolled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stabilization + Classic Pain Neuroscience Education (Experimental): Individuals in this group will undergo classical pain education (based on visual presentation or face-to-face instruction) along with core stabilization exercises targeting the muscles surrounding the spine. The exercises will be organized according to protocols reported in the literature as safe and effective and will include the following elements:
  * Exercises that activate the transversus abdominis and multifidus muscles (e.g., abdominal bracing, bird-dog, plank, side bridge)
  * Posture and spinal control exercises
  * Stretching and mobilization movements (lumbar flexion/extension, hip flexor stretches)
  * Each exercise will be performed in 2-3 sets of 10-15 repetitions, with the load increased according to participant tolerance.
  During the application process, participants will be provided with classic educational materials (e.g., verbal explanations or informative brochures) about the physiological basis of pain, movement safety, and exercise-related pain management. Thi
  Interventions: Other: Core Stabilization Exercises; Other: Classic Pain Neuroscience Education
- Core Stabilization + Virtual Reality-Assisted Pain Neuroscience Education (Experimental): Individuals in this group will receive SG-supported pain education in addition to the Group 1 protocol. Program details:
  1. Initial Session (Week 1)
     * 20-30 minutes of pain education modules in the SG environment
     * Information on the neurophysiological basis of pain, catastrophizing, and fear-avoidance behaviors
     * Reinforcement with interactive questions and short exercises
  2. Weekly Reinforcement (Weeks 2-6)
     * 10-15 minutes of short SG modules each week
     * Integration with core exercise sessions
  Interventions: Other: Core Stabilization Exercises; Other: Virtual Reality-supported pain neuroscience education program

INTERVENTIONS:
Other: Core Stabilization Exercises — Individuals in this group will undergo classical pain education (based on visual presentation or face-to-face instruction) along with core stabilization exercises targeting the muscles surrounding the spine. The exercises will be organized according to protocols reported in the literature as safe and effective and will include the following elements:
  * Exercises that activate the transversus abdominis and multifidus muscles (e.g., abdominal bracing, bird-dog, plank, side bridge)
  * Posture and spinal control exercises
  * Stretching and mobilization movements (lumbar flexion/extension, hip flexor stretches)
  * Each exercise will be performed in 2-3 sets of 10-15 repetitions, with the load increased according to participant tolerance.
Other: Classic Pain Neuroscience Education — During the application process, participants will be provided with traditional educational materials (e.g., verbal explanations or informational brochures) on the physiological basis of pain, movement safety, and pain management related to exercise. This training will not include virtual reality support.
  Arms: Core Stabilization + Classic Pain Neuroscience Education
Other: Virtual Reality-supported pain neuroscience education program — Details of the Virtual Reality-supported pain neuroscience education program:
  1. Introductory Session (Week 1)
     * 20-30 minutes of pain education modules in the VR environment
     * Information on the neurophysiological basis of pain, catastrophizing, and fear-avoidance behaviors
     * Reinforcement with interactive questions and short exercises
  2. Weekly Reinforcement (Weeks 2-6)
     * 10-15 minutes of short VR modules each week
     * Integration with core exercise sessions
  Arms: Core Stabilization + Virtual Reality-Assisted Pain Neuroscience Education

SUMMARY:
Chronic nonspecific low back pain is a multifactorial condition involving not only biomechanical but also psychological and neurocognitive components, in which factors such as kinesiophobia and pain catastrophizing contribute to pain persistence and disability. Pain Neuroscience Education (PNE) aims to reconceptualize pain, reduce fear-avoidance behaviors, and improve function, particularly when combined with exercise, although traditional educational methods may be limited in explaining abstract concepts. Virtual reality (VR) offers an interactive and engaging platform that may enhance the effectiveness of PNE by facilitating cognitive restructuring and increasing motivation, with evidence of short-term benefits on pain and kinesiophobia. Integrating VR-supported PNE with core stabilization exercises may simultaneously address biomechanical and cognitive processes, thereby providing a more comprehensive rehabilitation approach. Accordingly, this study aims to examine the effects of adding VR-supported pain education to core stabilization exercises on pain, kinesiophobia, pain catastrophizing, functional status, and balance in individuals with chronic nonspecific low back pain.

DETAILED DESCRIPTION:
Chronic nonspecific low back pain (CNSLBP) is a complex condition that cannot be explained solely by biomechanical factors and also involves psychological and neurocognitive components. Kinesiophobia, pain catastrophizing, and maladaptive pain beliefs have been shown to play a significant role in the chronification of pain and the increase in disability. Therefore, the Pain Neuroscience Education (PNE) approach, which focuses on the neurophysiology of pain, helps individuals reconceptualize pain, reduces fear-avoidance behaviors, and supports functional improvement. When applied in combination with exercise, PNE has been reported to provide additional benefits in reducing pain intensity, kinesiophobia, and catastrophizing. However, conventional educational methods may be limited in conveying abstract neurophysiological concepts.

At this point, virtual reality (VR) technology may enhance the effectiveness of pain education by providing an interactive and engaging learning environment. VR has been reported to facilitate cognitive restructuring in individuals with chronic pain and to increase motivation for participation. Moreover, VR-supported rehabilitation interventions have been shown to have short-term positive effects on pain and kinesiophobia in chronic pain conditions.

Core stabilization exercises are an effective method for improving postural control and functional stability in low back pain by regulating the activation of muscles surrounding the spine. However, purely physical approaches may be insufficient in adequately addressing the psychological dimensions of pain. Integrating VR-supported PNE into an exercise program may broaden the scope of rehabilitation by simultaneously influencing both biomechanical and cognitive processes. Therefore, this study aims to investigate the effects of adding VR-supported pain education to core stabilization exercises on pain, kinesiophobia, pain catastrophizing, functional status, and balance in individuals with CNSLBP. This holistic approach is expected to provide an innovative contribution to conventional exercise protocols and to shed light on the biopsychosocial management of chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 65
* Have a diagnosis of nonspecific low back pain with a history of low back pain lasting at least 3 months
* Have no specific pathologies that could cause low back pain (e.g., tumor, infection, fracture, inflammatory disease)
* Be able to walk independently and have the capacity to exercise
* Mini Mental State Examination score >23

Exclusion Criteria:

* Individuals who have undergone lumbar surgery within the last year,
* Individuals with central or peripheral neurological disorders (e.g., multiple sclerosis, peripheral neuropathy, Parkinson's disease),
* Those with vestibular, visual, or balance disorders (those at risk of dizziness or nausea during virtual reality applications),
* Those with serious cardiopulmonary or systemic diseases,
* Those with psychiatric disorders or a diagnosis of severe depression, those who are pregnant
* Individuals with a history of dizziness, epilepsy, or visual disturbances associated with virtual reality use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Severity of Pain | 6 week
  A visual analog scale will be used to assess patients' current pain intensity. This scale is one of the most commonly used scales for assessing pain intensity during rest, activity, and at night. The scale features a 10 cm line on which the patient can mark their pain intensity. Patients are asked to indicate the degree of their pain intensity on the line, ranging from no pain (left side) to unbearable pain (right side).
Functional Status | 6 week
  The level of disability resulting from low back pain will be assessed using the Oswestry Disability Index (ODI). The ODI was developed by Fairbank et al. in 1980, and its Turkish validity and reliability were established by Yakut et al. The ODI is one of the most widely used instruments for determining the extent to which daily living activities and functional status are affected by pain in individuals with low back pain.

SECONDARY OUTCOMES:
Balance | 6 week
  To determine the balance level of individuals with CNSLBP, the Biodex Balance System, which has been reported to be a reliable and valid assessment tool, will be used. Balance assessment on the Biodex Balance System is performed separately under dynamic and static conditions. The system consists of a balance platform that can tilt up to approximately 20° and has a 360° range of motion. The platform moves in the mediolateral (M-L) and anteroposterior (A-P) directions. Under dynamic conditions, the device calculates the degree of platform tilt, whereas under static conditions it measures deviations of the center of pressure. The difficulty level of the test is adjusted by changing the surface stability of the platform. On the balance platform, stability levels range from 12 (minimum stability) to 0 (maximum stability). In this study, the surface stability was set at Level 6. The Biodex Balance System quantifies balance loss using the average of the M-L and A-P scores, with higher scores
Pain Catastrophizing | 6 week
  The Pain Catastrophizing Scale (PCS) is a 13-item questionnaire designed to assess the extent of catastrophic thoughts and feelings related to pain in individuals experiencing pain. Each item is rated on a 5-point scale, with higher scores indicating greater levels of catastrophizing. Subscale scores are calculated by summing the scores of the corresponding items, and the total score is obtained by summing all items. PCS scores range from 0 to 52.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Merkez, Kirşehi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No